CLINICAL TRIAL: NCT05278312
Title: Measuring the Effect of Using the Arabic Otago Exercise Program on Falls and Falls-related Outcomes in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alia A. Alghwiri, Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/2021/9426
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Older Adults
Keywords: Otago Exercise Program; Falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): Older adults will receive the Otago Exercise Program for 8 weeks plus health awareness videos.
  Interventions: Other: Otago Exercise Program
- Control group (No Intervention): Older adults will receive only health awareness videos every 2 weeks.

INTERVENTIONS:
Other: Otago Exercise Program — A Home-based Exercise Program to improve strength and balance and prevent falls.
  Arms: Otago Exercise Program

SUMMARY:
Falls are common in older adults and may lead to disability or even death. Therefore, exercise programs that focus on preventing falls by improving strength and balance are important to investigate in older adults. One of the home-based exercise programs that was found effective in reducing the risk of falling and the rate of subsequent falls in older adults is the Otago exercise program (OEP). The OEP is an individualized home based retraining program that works mainly on balance and lower extremity strength through several progressive resistive exercises.

Therefore, this study aims to assess the effectiveness of this program on falls prevention and falls-related outcomes using a Randomized Controlled Trial in a sample of Jordanian older adults.

DETAILED DESCRIPTION:
❖ Research ethics: This study got the ethics approval from the IRB at Jordan University Hospital at University of Jordan. A consent form that contains the study procedures will be prepared and signed from all participants. To insure the privacy of participants, every older adult will be assigned a study identification number. All results will be stored in a locked cabinet/computer only accessible by the researchers.

❖ Participants: Data will be collected prospectively from older adults in Jordan. Older adults will be approached to complete the program via Jordan University Hospital, community based organizations (e.g. Help-Age International Jordan) and social media platforms such as Facebook and WhatsApp.

❖ Design:

● This will be a single blinded randomized controlled trial study with 2 groups: treatment group who will receive the OEP plus health awareness videos every 2 weeks and a control group who will receive the same health awareness videos only every 2 weeks.

1. Eligible older adults will be recruited for the RCT.
2. Baseline assessment will be conducted by a blind assessor.
3. Participant will be randomized using a computer-based randomization tool into either the treatment (OEP) or the control group (awareness videos). The treatment group will receive the OEP for 8 weeks plus health awareness videos. The control group will receive the same health awareness videos every 2 weeks for 8 weeks. The treatment group will be trained by a researcher different from the one conducting the assessments.

The following topics will be covered in the health awareness videos:

* Be physically active.
* Maintain healthy bones, joints and muscles.
* Combat depression.
* Sleep.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are 60 years of age and older.
* Who can read and write in Arabic language.
* Who are able to walk outdoors with no more support than a single point cane.

Exclusion Criteria:

* Who have a serious orthopedic condition (e.g., recent lower limb surgery, severe arthritis of a lower limb) or major neurological disorder (e.g., stroke with unilateral or bilateral paresis, Parkinson disease or multiple sclerosis) that could restrict functional mobility.
* Who are unable to comprehend study information and consent processes due to any illness including dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of falls | 2 months post intervention.
  The effect of the intervention on the incidence of falls.
Incidence of falls | 6 months post intervention.
  The effect of the intervention on the incidence of falls.
Incidence of falls | 12 months post intervention.
  The effect of the intervention on the incidence of falls.

SECONDARY OUTCOMES:
Fear of Falling (using the Falls Efficacy Scale-International) | 2 months post intervention.
  The effect of the intervention on fear of falling. The total score ranges between 16 and 64 with a higher score indicates greater fear of falling (worse).
Balance (using Chair balance test and Four test balance scale) | 2 months post intervention.
  The effect of the intervention on balance. The time taken to conduct these balance tasks are timed using a stopwatch. The longer the time taken by the participant to perform the tasks, the worse the balance. There is no minimum or maximum scores for these tests.
Mobility (using Timed-Up and go) | 2 months post intervention.
  The effect of the intervention on mobility. This assessments of mobility is timed out using a stopwatch.
Muscle strength (Hand grip and Quadriceps muscle strength using a dynamometer) | 2 months post intervention.
  The effect of the intervention on upper and lower extremity muscle strength. The strength of Hand grip and Quadriceps muscle will be assessed using a dynamometer in kilograms.
The Quality of sleep (Using Pittsburgh Sleep Quality Index) | 2 months post intervention.
  The effect of the intervention on the Quality of sleep. The total score ranges from 0 to 21 with a higher score indicates poor quality of sleep (worse).
the severity of Anxiety and Depression (using Hospital Anxiety and Depression Scale) | 2 months post intervention.
  The effect of the intervention on the severity of Anxiety and Depression. The total score for each subscale of the HADS ranges from 0 to 21 with higher score indicates more severe anxiety or depression (worse).
The Quality of Life (using Medical Outcomes Study Short Form 12) | 2 months post intervention.
  The effect of the intervention on Quality of Life. The total score ranges between 0% to 100% with higher score indicates a better quality of life (better).
Cognitive ability (using Montreal Cognitive Assessment) | 2 months post intervention.
  The effect of the intervention on Cognitive ability. The total score ranges from 0 to 30 points with a score of 25 or less indicating cognitive impairment (worse).
Sarcopenia (using the bio-impedance analysis) | 2 months post intervention.
  The effect of the intervention on muscle mass. Muscle mass will be measured using a bio-impedance analysis device (InBody).
Pain (using pain rating scale) | 2 months post intervention.
  The effect of the intervention on pain. The total score of PRS ranges between 0 to 10 with higher score indicates more pain and interference with discomfort (worse).
Activities of daily living (using Katz index of daily living) | 2 months post intervention.
  The effect of the intervention on independence in performing activities of daily living. The total score ranges between 0 to 6 with higher score indicates a better independence.

CONTACTS AND LOCATIONS:
Overall Officials: Alia A. Alghwiri, PhD, Principal Investigator — University of Jordan
Locations (2):
- Jordan (2):
  - Alia Alghwiri, Amman
  - University of Jordan, Amman

IPD SHARING:
Plan to Share IPD: No